CLINICAL TRIAL: NCT01963156
Title: Synchronization to Improve Non-Adherence to Cardiovascular Medications (SyNCMed)
Brief Title: Synchronization to Improve Non-Adherence to Cardiovascular Medications
Acronym: SyNCMed
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: CVS Caremark (Industry)
Responsible Party: Principal Investigator, Niteesh K. Choudhry, MD, PhD, Associate Professor, Harvard Medical School, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00008813
Record Dates: First submitted 2013-10-10; First posted 2013-10-16 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Disease; Cardiovascular Disease; Diabetes Mellitus
Keywords: Prescription synchronization; Cardiovascular disease; Medication adherence; Randomized controlled trial; Chronic disease; Pharmacy benefit design; Quality improvement
MeSH Terms: conditions — Chronic Disease; Cardiovascular Diseases; Diabetes Mellitus; Medication Adherence

ARMS (2):
- Prescription synchronization (Experimental)
  Interventions: Behavioral: Prescription synchronization
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Prescription synchronization — Each patient's medication that has the greatest quantity of pills on hand after randomization will be defined as the "index "medication and partial supplies will be provided for all other eligible medications in order to synchronize all of a patient's medication. Prescribers will be contacted for a new prescription to ensure all eligible medications are on the same renewal schedule.
  Randomization will occur within strata of whether patients are enrolled in the "ReadyFill@Mail" program. Once synchronized, patients who are not enrolled in the ReadyFill@Mail program will initiate their own refills. Patients who are enrolled in the ReadyFill@Mail program will have their refills automatically filled, however patients may disenroll from ReadyFill@Mail at any time, in which case they will initiate their own refills. Patients may disenroll in whole or in part from the program at any point.
  Arms: Prescription synchronization

SUMMARY:
The aim of this study is to evaluate if synchronizing when patients with diabetes and/or coronary artery disease fill their prescriptions improves long-term adherence to these medications.

ELIGIBILITY:
We will enroll patients 18 years of age and older who within 6 months of study enrollment have filled ≥ 2 medications intended for long-term use (i.e. maintenance medications) by mail order at CVS Caremark. At least 1 of these 2 medications of must be for the treatment of diabetes or cardiovascular disease. In addition, these medications must be delivered on two or more unique delivery dates, there must be at least one refill remaining for all eligible medications and either all or none of their prescriptions must be enrolled in the ReadyFill@Mail program (see Intervention Description for details).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3675 (Actual)
Dates: Start 2013-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Medication adherence | 12 months
  Average adherence to medications for the treatment of cardiovascular disease and diabetes medications as assessed using administrative pharmacy claims

SECONDARY OUTCOMES:
Full adherence to medications for the treatment of diabetes or cardiovascular disease | 12 months
  Percent of subjects achieving full adherence (defined as a Medication Possession Ratio > 80%) to medications for cardiovascular disease and diabetes

OTHER OUTCOMES:
Rates of de-synchronization | 12 months
  Rate at which members whose prescriptions have been synchronized elect to discontinue with the synchronization during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Niteesh K Choudhry, MD, PhD, Principal Investigator — Brigham and Women's Hospital/Harvard Medical School
Locations (1):
- CVS Caremark, Woonsocket, Rhode Island, United States